CLINICAL TRIAL: NCT05656963
Title: Influence Factors and Preliminary Mechanism of High Incidence of Thrombotic Events in Patients With Idiopathic Membranous Nephropathy and Diabetes Kidney Disease
Brief Title: The Influencing Factors and Mechanism of High Incidence of Thrombotic Events in Patients With MN and DKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yipeng Liu (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(102)
Record Dates: First submitted 2022-11-24; First posted 2022-12-20 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Glomerulonephritis, Membranous; Diabetic Nephropathies; Thrombelastography; Thromboembolism
MeSH Terms: conditions — Glomerulonephritis, Membranous; Diabetic Nephropathies; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic membranous nephropathy: Patients with idiopathic membranous nephropathy proved by renal biopsy
  Interventions: Other: Grouping based on previous laboratory results, no intervention.
- Non-Idiopathic membranous nephropathy: Other primary glomerular diseases except membranous nephropathy
  Interventions: Other: Grouping based on previous laboratory results, no intervention.
- Diabetic kidney disease: Patients with clinical diagnosis of diabetes and kidney disease
  Interventions: Other: Grouping based on previous laboratory results, no intervention.

INTERVENTIONS:
Other: Grouping based on previous laboratory results, no intervention. — The patients were grouped according to the results of previous inpatient tests, and no intervention measures were taken.

SUMMARY:
Influence factors and preliminary mechanism of high incidence of thrombotic events in patients with idiopathic membranous nephropathy and diabetes kidney disease

DETAILED DESCRIPTION:
According to the results of renal biopsy, the patients were divided into three groups: membranous nephropathy group (MN), non-membranous nephropathy group (non-MN) and diabetes kidney disease group (DKD). Collect the basic data and TEG test results of the enrolled patients. (1) ① According to TEG results, the enrolled patients were divided into two groups: hypercoagulable group (CI > 3) and non-hypercoagulable group (CI ≤ 3). The basic data and related laboratory indicators of the two groups were compared - to explore the influencing factors of hypercoagulable (objective X); ② Compare the parameters related to TEG and coagulation routine between MN group and non-MN group, DKD group and non-MN group respectively - find out the coagulation index (target Y) of the difference between groups; ③ Build regression models for different target Y - explore the influencing factors of grouping variables (MN vs non MN or DKD vs non MN) on Y after adjusting other covariates; (2) ① According to whether the patients in the group had thrombotic events or not, all the patients in the group with thrombotic events were divided into MN thrombotic events group and non-MN thrombotic events group according to pathological diagnosis, and the TEG, coagulation and other related laboratory results and basic data between the two groups were compared (explore the unique factors and processes that affect the occurrence of thrombotic events in MN group compared with non-MN group); ② According to whether the patients in the MN group who were hospitalized for many times had thrombotic events, the patients were divided into the MN group with thrombotic events and the MN group without thrombotic events. The TEG, coagulation and other related laboratory results and basic data between the two groups were compared (to explore the factors and processes that affect the occurrence of thrombotic events in the MN group).

ELIGIBILITY:
Inclusion Criteria:

1. Primary glomerular disease patients with renal biopsy results (without hormone or immunosuppressive therapy) and patients with clinical diagnosis of diabetes kidney disease;
2. Age 18-70;
3. The liver function is normal.

Exclusion Criteria:

1. Other secondary kidney diseases except diabetes; Acute renal injury; Chronic kidney disease stage 5;
2. There are risk factors of hypercoagulability, such as acute infection, recent trauma, surgery or cancer, pregnancy;
3. Anticoagulant and antiplatelet drugs were given within one week;
4. Plasma infusion, plasma exchange or hemodialysis within one month;
5. There is a history of thrombotic disease or hemorrhagic disease before renal puncture;
6. Participated in other clinical studies within three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were diagnosed as primary glomerular disease by renal puncture biopsy and diabetes renal disease by clinical diagnosis and underwent thromboelastography (TEG) examination at the same time were newly treated patients and were not treated with hormone and other immunosuppressants.
Sampling Method: Non-Probability Sample
Enrollment: 741 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Factors influencing the high incidence of thrombotic events in patients with membranous nephropathy and diabetic nephropathy | 2021-2024
  Collect the basic data of the enrolled patients, including admission blood pressure, smoking, drinking history, the use of statins, anticoagulants and antiplatelet drugs, and blood test indicator. All indicators for inclusion in the analysis are presented in full by subgroup. ① the enrolled patients were divided into two groups according to TEG results: hypercoagulable group (CI > 3) vs non hypercoagulable group (CI ≤ 3). The basic data and related laboratory parameters of the two groups were compared to explore the influence of hypercoagulability factors (AIM X); ② Comparison of TEG and coagulation routine related parameters between MN and non MN group, DKD and non MN group - to find the coagulation indexes (target Y) that differ in TEG and coagulation routine between groups; ③ Regression models were constructed separately for different targets Y - to explore the influence of grouping variables (MN vs non MN or DKD vs non MN) on y after adjusting for other covariates;
Specific link between high incidence of thrombotic events in patients with membranous nephropathy and diabetic nephropathy | 2021-2024
  ① Based on collecting whether all the patients enrolled in multiple hospitalizations had thrombotic events, all the patients enrolled with thrombotic events were divided into MN with thrombotic events group and non MN with thrombotic events group according to the pathological diagnosis, and relevant assay results such as TEG, coagulation and basic data were compared between the two groups (to explore the specific factors and processes influencing the occurrence of thrombotic events specifically in the MN group compared to the non MN group); ② Based on whether thrombotic events occurred in patients within the Mn group enrolled in multiple hospitalizations, patients were divided into Mn with thrombotic events and Mn without thrombotic events groups, and relevant laboratory results and basic data such as TEG and coagulation were compared between the two groups (to explore factors and processes influencing the occurrence of thrombotic events in patients within the MN group).

CONTACTS AND LOCATIONS:
Overall Officials: Yipeng Liu, Study Chair — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No